CLINICAL TRIAL: NCT00077194
Title: A Phase II Study Of Depsipeptide, A Histone Deacetylase Inhibitor, In Relapsed Or Refractory Mantle Cell Or Diffuse Large Cell Non-Hodgkin's Lymphoma
Brief Title: FR901228 in Treating Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02571; MAYO-MC0287; NCI-5961; CDR0000349660 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-02-10; First posted 2004-02-11 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2005-02

CONDITIONS: Lymphoma
Keywords: recurrent adult diffuse large cell lymphoma; recurrent mantle cell lymphoma; recurrent adult Burkitt lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Burkitt Lymphoma | interventions — romidepsin

ARMS (1):
- Arm I (Experimental): Patients receive FR901228 (depsipeptide) IV over 4 hours on days 1, 8, and 15. Treatment repeats every 28 days for at least 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: romidepsin

INTERVENTIONS:
Drug: romidepsin

SUMMARY:
This phase II trial is studying how well FR901228 works in treating patients with relapsed or refractory non-Hodgkin's lymphoma. Drugs used in chemotherapy, such as FR901228, work in different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the response rate (complete and partial) in patients with relapsed or refractory Burkitt's, mantle cell or diffuse large cell non-Hodgkin's lymphoma treated with FR901228 (depsipeptide).

II. Determine the safety and feasibility of this drug, in terms of incidence and maximum grade of toxicity and courses delayed or doses reduced, in these patients.

III. Determine the 2-year progression-free survival and overall survival of patients treated with this drug.

IV. Correlate tumor expression of BCL-2, BCL-6, BAX, and RAS with response in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive FR901228 (depsipeptide) IV over 4 hours on days 1, 8, and 15. Treatment repeats every 28 days for at least 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months until disease progression and then every 6 months until 5 years from study registration.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed aggressive B-cell non-Hodgkin's lymphoma of 1 of the following cellular types:

  * Diffuse large cell
  * Mantle cell
  * Burkitt's
* Relapsed or refractory disease

  * No more than 2 prior regimen for patients with refractory disease
  * Any number of prior therapies (including peripheral blood stem cell or bone marrow transplantation) allowed for patients with relapsed disease provided there was an objective response to the most recent therapy
* Measurable disease

  * At least 1 lesion ≥ 1.5 cm in diameter
* No transformed lymphoma
* No CNS lymphoma
* Ineligible for, refused, or relapsed after stem cell transplantation

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Hematopoietic

* Absolute neutrophil count ≥ 1,000/mm^3 (500/mm^3 in patients with extensive bone marrow involvement [> 50%] or hypersplenism with palpable splenomegaly)
* Platelet count ≥ 75,000/mm^3 (50,000/mm^3 in patients with extensive bone marrow involvement or hypersplenism with palpable splenomegaly)

Hepatic

* Bilirubin ≤ upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2 times ULN
* AST ≤ 2 times ULN

Renal

* Creatinine ≤ ULN

Cardiovascular

* QTc < 500 msec by ECG
* Cardiac function ≥ 50% by MUGA
* No prior serious ventricular arrhythmia
* No New York Heart Association class III or IV congestive heart failure
* No significant cardiac hypertrophy by ECG
* No other significant cardiac disease

Pulmonary

* No chronic obstructive pulmonary disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No active infection
* No diabetes
* No other uncontrolled serious medical condition

PRIOR CONCURRENT THERAPY:

Chemotherapy

* Prior cumulative doxorubicin dose < 450 mg/m^2
* Prior cumulative mitoxantrone dose < 112 mg/m^2
* Prior doxorubicin equivalent dose < 450 mg/m^2 (for patients who have previously received both doxorubicin and mitoxantrone)

Other

* Recovered from all prior therapy
* No prior histone deacetylase inhibitor therapy
* No concurrent medication associated with QTc prolongation, such as dolasetron
* Concurrent hydrochlorothiazide, furosemide, or other diuretics allowed provided patient is on concurrent potassium chloride supplementation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2004-01; Primary Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy L. Bartlett, MD, Study Chair — Washington University Siteman Cancer Center
Locations (4):
- United States (4):
  - Howard University Cancer Center at Howard University Hospital, Washington D.C., District of Columbia
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin